CLINICAL TRIAL: NCT06966765
Title: Accelerated vs Standard Approach to Continuous Veno-venous Hemodiafiltration Post-hemoperfusion (ASAP) in Severe Acute Diquat Poisoning: a Multi-center, Cluster, Randomized, Controlled Trial
Brief Title: Accelerated vs Standard Approach to Continuous Veno-venous Hemodiafiltration Post-hemoperfusion (ASAP) in Severe Acute Diquat Poisoning
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Hao Sun, Principal Investigator, Clinical Associate Professor, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-12122-2
Record Dates: First submitted 2025-05-04; First posted 2025-05-13 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Diquat Poisoning
Keywords: diquat; continuous kidney replacement therapy
MeSH Terms: interventions — Continuous Renal Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Accelerated Initiation (Experimental): Participants in this experimental arm will receive CVVHDF within 12 hours of eligibility confirmation. This 12-hour window includes the time required to obtain consent, place a dialysis catheter, and initiate CVVHDF.
  Interventions: Procedure: Continuous Veno-Venous Hemodiafiltration
- Standard Initiation (Active Comparator): Treating clinician(s) will not be encouraged to initiate CVVHDF unless the patient develops AKI, defined by any of the following criteria, according to the Kidney Disease: Improving Global Outcomes (KDIGO) guidelines. CVVHDF may be initiated at any time at the discretion of the treating clinician(s). However, if CVVHDF is initiated without the participant meeting AKI diagnostic criteria, treating clinician(s) will be asked to document the primary rationale. Conversely, even when AKI criteria are met, there is no obligation to initiate CVVHDF if the treating clinician(s) judge that alternative medical interventions are more appropriate based on current standard care; in such cases, the reasons for withholding CVVHDF should also be documented.
  Interventions: Procedure: Continuous Veno-Venous Hemodiafiltration

INTERVENTIONS:
Procedure: Continuous Veno-Venous Hemodiafiltration — CVVHDF will be delivered following hemoperfusion with a dialysate-to-replacement fluid ratio maintained at 1:1, a blood flow rate of 150-200 mL/min, and a target dialysis dose of 30 mL/kg/h (excluding additional fluid removal). Regional anticoagulation (e.g., heparin or other agent per device requirements) will be used to prevent clotting within the circuit. Once CVVHDF is initiated in either arm, it will not be discontinued until one of the following encountered: (i) death; or (ii) a change in goals of care with withdrawal of life-sustaining interventions; or (3) recovery of kidney function, as determined by treating clinician(s), such that CVVHDF will be no longer required. However, CVVHDF will be reinitiated at the discretion of treating clinician(s), if kidney function comes suboptimal after a period of discontinuation.

SUMMARY:
Diquat (1,1'-ethylene-2,2'-bipyridinium) is a bipyridine herbicide that shares a similar physicochemical structure and redox cycling mechanism with paraquat. Upon ingestion, it is rapidly absorbed and distributed to the gastrointestinal tract, kidneys, liver, skeletal muscle, lungs, myocardium, and central nervous system. Patients with severe diquat poisoning often develop toxic encephalopathy, circulatory collapse, and multi-organ dysfunction. Extracorporeal treatments, including hemoperfusion, hemodialysis, and continuous kidney replacement therapy (CKRT), are widely employed to manage diquat poisoning. Continuous veno-venous hemodiafiltration (CVVHDF), the most frequently used CKRT modality, is primarily indicated for acute kidney injury (AKI). AKI occurs in up to 73.3% of patients with acute diquat poisoning, and nearly all patients with severe acute diquat poisoning are at risk of developing AKI. In clinical practice, patients with severe acute diquat poisoning are typically defined as those with a plasma diquat concentration of ≥1000 ng/mL measured at the time of presentation to the emergency department (ED). However, the Extracorporeal Treatments in Poisoning (EXTRIP) workgroup has not issued any definitive recommendations on initiating extracorporeal treatments for diquat poisoning, and the optimal timing for starting CVVHDF has yet to be evaluated in clinical trials. Currently, the standard practice delays initiation of CVVHDF until AKI has developed. Accordingly, this study proposes a pragmatic cluster-randomized controlled trial (RCT) to determine whether, in severe acute diquat poisoning patients, accelerated initiation of CVVHDF following hemoperfusion is preferred compared to a standard approach in which CVVHDF is initiated only in the presence of AKI or at the discretion of the treating clinician.

ELIGIBILITY:
Inclusion criteria:

1. Age ≥ 18 years; and
2. A history of oral exposure to diquat solution, reported by patient(s) or their legal proxies; and
3. An exposure time (time form exposure to presentation at ED) ≤ 48 hours, reported by patient(s) or their legal proxies; and
4. Plasma diquat concentration measured upon ED presentation ≥ 1,000 ng/mL.

Exclusion criteria:

1. Evidence of co-ingestion of other toxic substances alongside diquat; and/or
2. Withholding of CVVHDF due to limitations on the escalation of life-sustaining therapies; and/or
3. Any CKRT within the previous 2 months; and/or
4. Kidney transplant within the past 365 days; and/or
5. Known pre-hospitalization advanced chronic kidney disease, defined by an estimated glomerular filtration rate calculated using serum creatine (eGFRer) of less than 30 mL/min/1.73 m2 by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation, if pre-hospitalization serum creatine is available; and/or (6) Treating clinician(s) believe(s) that either immediate or deferral of CVVHDF initiation is mandated; and/or (7) Pregnant or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Estimated)
Dates: Start 2027-01-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality rate | 90 days within the index date of randomization
Time from exposure to death | 90 days within the index date of randomization
  The primary outcome measure included time from exposure to death.

SECONDARY OUTCOMES:
ICU-free days | 90 days within the index date of randomization
Ventilator-free days | 90 days within the index date of randomization
Vasoactive-free days | 90 days within the index date of randomization
CVVHDF dependence rate | 90 days within the index date of randomization
Hospitalization-free days | 90 days within the index date of randomization
Major adverse kidney events rate | 90 days within the index date of randomization
  The secondary outcome measure included major adverse kidney events at 90 days after randomization, defined as the composite of death, CVVHDF dependence, or sustained reduction of kidney function (defined as eGFR <75% of the lowest eGFR measured during hospitalization).